CLINICAL TRIAL: NCT02907203
Title: Clinical Investigation of the GORE® Drug-Coated PTA Balloon Catheter (GORE® DCB Catheter) for Conformité Européene (CE) Mark Approval
Brief Title: Clinical Investigation of the GORE® Drug-Coated PTA Balloon Catheter (GORE® DCB Catheter)
Acronym: DCB
Status: Completed | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCB 15-02
Record Dates: First submitted 2016-09-12; First posted 2016-09-20 (Estimated); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: PAD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | Unapproved Device: Yes

ARMS (1):
- Drug Coated Balloon (Experimental): Prospective, multi-center, single-arm study characterizing outcomes in subjects with Peripheral Artery Disease (PAD) lesions treated with percutaneous transluminal angioplasty (PTA) using the GORE® DCB Catheter.
  Interventions: Device: Drug Coated Balloon

INTERVENTIONS:
Device: Drug Coated Balloon — Prospective, multi-center, single-arm study characterizing outcomes in subjects with Peripheral Artery Disease (PAD) lesions treated with percutaneous transluminal angioplasty (PTA) using the GORE® DCB Catheter.

SUMMARY:
This study will assess the safety and performance of the Gore drug-coated balloon in the treatment of de novo and restenotic atherosclerotic lesions in the superficial femoral and popliteal arteries of patients with symptomatic PAD.

DETAILED DESCRIPTION:
The primary objective of the clinical investigation is to evaluate the safety and performance of the Gore drug-coated balloon in the treatment of de novo and restenotic atherosclerotic lesions in the superficial femoral and popliteal arteries (SFA/PA) of patients with symptomatic PAD.

The performance of the GORE® DCB Catheter is superior to a performance goal derived from literature reports of uncoated PTA balloons, measured six months after intervention.

ELIGIBILITY:
Inclusion Criteria:

* PAD patients with Rutherford Class 2 - 4
* De novo or restenotic lesions, including total occlusions of the SFA/PA
* 1 lesion which may include one or more regions of luminal narrowing ≥70% with a total combined lesion length between 30 - 150mm and a reference vessel diameter of 4 - 6mm
* 1 patent tibial or peroneal artery

Exclusion Criteria:

* Surgical or endovascular access in the Target limb/vessel within the previous 30 days
* Prior treatment of the Target lesion with PTA within 90 days or any prior treatment with drug-coated balloon
* Prior treatment of the Target vessel with stenting or bypass
* Iliac artery inflow lesions that cannot be successfully treated during the Index procedure
* Acute or subacute thrombus or arterial aneurysm in Target limb
* Severe calcification that renders the Target lesion non-dilatable
* Acute or chronic renal dysfunction (serum creatinine ≥2.5 mg/dL)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitats - Herzzentrum Freiburg, Bad Krozingen, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug Coated Balloon
Started | 52
Completed | 44
Not Completed | 8
Not completed — Death | 1
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 3
Not completed — Surgical bypass | 1

BASELINE CHARACTERISTICS:
Arm/Group | Drug Coated Balloon
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 52
Mean Lesion Diameter Post Procedure(mm) [Mean (Standard Deviation); unit: milimeters] — The lesion diameter at the completion of the procedure is used as baseline from which the loss was calculated at six months.
  milimeters | 4.01 (0.69)

OUTCOME MEASURES:

1. Primary Outcome: Late Lumen Loss (LLL)
Description: Six month late lumen loss (LLL) is defined as the difference in minimum lumen diameter of the Target lesion between the time points immediately post-intervention and the 6-month follow-up angiography or at the time of a Clinically Driven Target Lesion Revascularization (CD TLR), whichever is earlier.
Time Frame: Six months
Population: Of the 44 subjects completed the study, the late lumen loss was only available for 37 subjects, rest were treated as missing data.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Drug Coated Balloon
Number analyzed (Participants) | 37
mm | -0.17 (0.98)
Statistical Analysis 1: Comparison: Drug Coated Balloon; Test type: Non-Inferiority — Compared with the Performance Goal: 0.9mm; p = 0.000, t-test, 2 sided; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.5 to 0.152], Standard Deviation 0.98

2. Secondary Outcome: Number of Subjects With Freedom From Major Adverse Events
Description: A composite 30-day safety endpoint of freedom from Major Adverse Events (MAE), defined as i) death, ii) Clinically-Driven Target Vessel Revascularization (CD TVR), or iii) amputation above the metatarsals, resulting from a vascular event, in the treated leg (Target limb amputation).
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Coated Balloon
Number analyzed (Participants) | 52
Participants | 52

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | Drug Coated Balloon
All-Cause Mortality (participants affected / at risk) | 1/52
Serious Adverse Events (participants affected / at risk) | 27/52
Other Adverse Events (participants affected / at risk) | 13/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Coated Balloon (N=52)
Coagulation disorder (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Coronary artery disease (Cardiac disorders) | 1 (1)
Mitral valve insufficiency (Cardiac disorders) | 1 (1)
Multiple vessel coronary artery disease (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Non STEMI (Cardiac disorders) | 1 (1)
Triple vessel disease (Cardiac disorders) | 1 (1)
Cataract (right) (Eye disorders) | 1 (1)
Esophagitis ulcerative (Gastrointestinal disorders) | 1 (1)
Aspiration pneumonia (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Perineal abscess (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Fracture of pelvis (Injury, poisoning and procedural complications) | 1 (2)
Fractured ribs (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture L3 (Injury, poisoning and procedural complications) | 1 (1)
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 2 (2)
Post angioplasty restenosis (Injury, poisoning and procedural complications) | 4 (4)
Second degree burns (Injury, poisoning and procedural complications) | 1 (1)
Shoulder fracture (Injury, poisoning and procedural complications) | 1 (1)
Superficial femoral arterial restenosis (Injury, poisoning and procedural complications) | 2 (2)
Diabetes mellitus aggravated (Metabolism and nutrition disorders) | 1 (1)
Limb hyperextension (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bleeding intracranial (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Nerve root impingement (Nervous system disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1)
Adventitial cystic disease (Vascular disorders) | 1 (1)
Femoral artery dissection (Vascular disorders) | 1 (1)
Femoral artery stenosis (Vascular disorders) | 2 (2)
Femoropopliteal stenosis (Vascular disorders) | 2 (2)
Hypertensive crisis (Vascular disorders) | 1 (2)
Iliac artery dissection (Vascular disorders) | 1 (1)
Iliac artery stenosis (Vascular disorders) | 2 (2)
Peripheral artery dissection (Vascular disorders) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 2 (2)
Peripheral artery stenosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug Coated Balloon (N=52)
Post angioplasty restenosis (Injury, poisoning and procedural complications) | 11 (11)
Superficial femoral arterial restenosis (Injury, poisoning and procedural complications) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT02907203/Prot_SAP_000.pdf